CLINICAL TRIAL: NCT04750993
Title: Comparison of the Frequency of Subclinic Synovitis in the Distal Interphalangeal Joints of the Hand in Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Lecturer Doctor, Ufuk University
Other Study IDs: 465/Gazi University
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis; Synovitis
MeSH Terms: conditions — Psoriasis; Synovitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: musculoskeletal ultrasonography — The presence of subclinic synovitis findings in the hand joints was evaluated with musculoskeletal ultrasonography.

SUMMARY:
In this cross-sectional study, it was planned to compare the frequency of subclinical synovitis in the distal interphalangeal joints of the hands in psoriasis patients. 28 patients followed up by the Dermatology Department with a diagnosis of psoriasis and referred to us and 28 healthy volunteers were included in the study. Participants' age, gender, body mass index (BMI), year of psoriasis diagnosis, treatments they received, and comorbid diseases were recorded as demographic information. Psoriasis Area and Severity Index (PASI) and Nail Psoriasis Severity Index (NAPSI) were calculated by a dermatologist.

Tenderness in the distal interphalangeal joints of both hands was evaluated by palpation.

Subsequently, the presence of ultrasonographic synovitis findings of the participants was examined by a physician who was experienced in musculoskeletal ultrasonography and was blind to clinical evaluations. Scoring was done with the EULAR GS / PD joint scoring system and EULAR-OMERACT composite scoring system. The scores of the most affected joint were used in statistical analysis. Comparisons were made between psoriasis and control groups in terms of scores. Relationships between variables in the psoriasis group were examined.

ELIGIBILITY:
Inclusion Criteria:

For patient group

1. Being over the age of 18
2. Being followed up by the Dermatology Department with a diagnosis of psoriasis and receiving topical or systemic treatment for this
3. Absence of clinically detected signs of arthritis
4. Absence of serious trauma, surgical intervention or injection in the joint areas to be evaluated.
5. Absence of any known inflammatory rheumatic disease For control group

1.> 18 years old 2. Absence of clinically detected signs of arthritis 3.Lack of clinical signs suggestive of psoriasis

Exclusion Criteria:

For patient group

1. To be <18 years old
2. Clinically detected evidence of arthritis
3. History of serious trauma, surgical intervention or injection in the joint areas to be evaluated
4. Having a known inflammatory rheumatic disease For control group

1. To be <18 years old 2. Having clinical signs suggestive of psoriasis 3. Having clinically detectable signs of arthritis 4. History of known inflammatory disease, severe trauma in the joint areas to be evaluated, surgical intervention, injection

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 psoriasis patients and 30 healthy volunteers were included in the study.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
GS/PD score | 8 month
  Intaarticular fluid (0 = absent, 1 = present), synovial hypertrophy (0 = absent, 1 = mild, 2 = moderate, 3 = severe), bone erosion (0 = absent, 1 = 2 erosion, 2 = More than 2 erosion), surrounding soft tissue swelling (0 = absent, 1 = mild, 2 = moderate) with gray scale; the presence of blood flow in the area with synovial proliferation with power Doppler (0 = no signal, 1 = less signal in one vessel, 2 = moderate signal at vascular intersections, 3 = intense signal on more than half of the joint surface) are evaluated and scored. GS and PD scores of the joint with the greatest involvement are used in statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No